CLINICAL TRIAL: NCT07134894
Title: Intensive Bimanual Therapy Versus Conventional Physical Therapy in Quadriplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Shareen Mehak, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0052
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Quadriplegic Cerebral Palsy; Cerebral Palsy (CP)
Keywords: Cerebral Palsy; Quadriplegic CP; Conventional Physical Therapy; Bimanual Coordination; Intensive Bimanual Therapy; Neuroplasticity; Task-Specific Training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Bimanual Therapy plus Conventional Physical Therapy (Experimental): Participants in this arm will receive a combination of Intensive Bimanual Therapy (IBT) and Conventional Physical Therapy (CPT) for 8 weeks. Therapy will be delivered three times per week, with two supervised sessions and one home-based session. Each 60-minute session will consist of 30 minutes of CPT-focusing on upper limb range of motion, strengthening, balance, and mobility-and 30 minutes of IBT, incorporating structured bimanual activities such as grasping, object transfer, buttoning, puzzle assembly, water pouring, and feeding with utensils. Activities will progress in complexity every two weeks, with parental guidance provided for home-based practice.
  Interventions: Behavioral: Intensive Bimanual Therapy plus Conventional Physical Therapy
- Conventional Physical Therapy Only (Active Comparator): Participants in this arm will receive Conventional Physical Therapy (CPT) for 8 weeks, delivered three times per week, with two supervised sessions and one home-based session. Each 40-minute session will include upper limb range of motion exercises, strengthening activities, and gross motor training, incorporating movements such as crawling, assisted stretches, squats, heel raises, step-ups, and knee lifts. Additional activities such as yoga-based poses, animal walks, single-leg stance, and stair climbing will be included to promote flexibility, balance, and functional mobility. The program focuses on general upper and lower limb conditioning without targeted bimanual coordination training.
  Interventions: Behavioral: Conventional Physical Therapy

INTERVENTIONS:
Behavioral: Intensive Bimanual Therapy plus Conventional Physical Therapy — A combined rehabilitation program delivered over 8 weeks, three sessions per week. Each 60-minute session includes 30 minutes of Conventional Physical Therapy (CPT) to improve range of motion, muscle strength, balance, and gross motor function, and 30 minutes of Intensive Bimanual Therapy (IBT) to enhance bilateral hand coordination and functional independence. IBT tasks progress from basic grasping and object transfer to complex daily activities such as buttoning, puzzle assembly, water pouring, and feeding with utensils. Two sessions are supervised by a physiotherapist and one is completed at home under caregiver guidance.
  Arms: Intensive Bimanual Therapy plus Conventional Physical Therapy
Behavioral: Conventional Physical Therapy — A standard physiotherapy program delivered over 8 weeks, three sessions per week, each lasting 40 minutes. Sessions focus on upper limb range of motion, strengthening, postural control, and functional mobility without targeted bimanual training. Exercises include assisted stretches, squats, heel raises, step-ups, knee lifts, yoga-based poses, animal walks, single-leg stance, and stair climbing to promote flexibility, balance, and gross motor performance. Two sessions are supervised by a physiotherapist and one is performed at home with caregiver supervision.
  Arms: Conventional Physical Therapy Only

SUMMARY:
Quadriplegic cerebral palsy (CP) is a severe neurological condition affecting motor control in all four limbs, often resulting in profound functional limitations in daily activities. Impaired upper limb function restricts children's ability to perform essential self-care, educational, and play tasks. Intensive Bimanual Therapy (IBT) is a rehabilitation approach that engages both hands in coordinated, repetitive, and task-specific activities to promote motor learning and functional independence. Conventional Physical Therapy (CPT), while widely used, primarily targets gross motor skills and may not fully address complex bilateral coordination needs.

This randomized controlled trial is designed to compare the effects of IBT and CPT on upper limb function in children with quadriplegic CP. Thirty children aged 2-6 years, classified at Gross Motor Function Classification System (GMFCS) levels III-IV, will be randomly assigned to either CPT alone or a combination of CPT and IBT. The Able Hand Questionnaire (ABL) will be used to measure functional bimanual use before and after an 8-week intervention period. The study aims to determine whether IBT offers additional benefits over standard therapy in enhancing bimanual coordination and functional independence in this population.

DETAILED DESCRIPTION:
Cerebral palsy is a non-progressive neurodevelopmental disorder caused by early brain injury, with quadriplegic CP representing one of the most severe forms. Children with this condition experience marked impairments in voluntary motor control, coordination, and postural stability. Functional use of the upper limbs is often significantly reduced, which impacts participation in self-care, education, and social activities.

Conventional Physical Therapy (CPT) typically focuses on improving gross motor performance, range of motion, strength, and mobility. While effective for some functional domains, it may not adequately target bilateral coordination, which is critical for everyday tasks. Intensive Bimanual Therapy (IBT) emphasizes the simultaneous use of both hands in structured, progressive, and meaningful activities such as dressing, feeding, and object manipulation. The intervention is based on neuroplasticity principles, incorporating high-repetition, task-specific practice, and active engagement to enhance motor control.

This study will be conducted at the University of Lahore Teaching Hospital. Eligible participants will be children aged 2-6 years with a diagnosis of quadriplegic CP, classified at GMFCS levels III-IV, with sufficient cognitive ability to follow simple instructions. Exclusion criteria include joint contractures limiting bimanual tasks, recent upper limb surgery, botulinum toxin injections within six months, or poor compliance potential.

Participants will be randomly allocated into two groups:

Group A (CPT only): Three 40-minute sessions per week for 8 weeks, including upper limb range of motion exercises, strengthening, balance activities, and functional mobility tasks.

Group B (CPT + IBT): Three 60-minute sessions per week for 8 weeks, combining CPT with 30 minutes of structured bimanual activities. These activities will progress from simple grasping and object transfer tasks to more complex functional activities such as buttoning, puzzle assembly, water pouring, and feeding with utensils. Home-based practice will be encouraged with parental guidance.

The primary outcome measure will be the Able Hand Questionnaire (ABL), which assesses functional use of the hands in daily activities. Assessments will be performed at baseline and after the 8-week intervention by a blinded assessor. Statistical analysis will be performed using non-parametric methods appropriate for the data distribution.

This trial is designed to provide evidence on whether the integration of IBT into standard therapy protocols can optimize functional upper limb outcomes for children with quadriplegic CP, ultimately informing best-practice rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Children with quadriplegic cerebral palsy.(Te Velde et al., 2021)
* The target population consisted of children aged 2-6 years (Horwood et al., 2019)
* Classified as level 3 and 4 in the GMFCS (Sogbossi et al., 2021)
* Muscle tone grade 2 at modified Ashwarth scale.(Sogbossi et al., 2021)
* Sufficient cognitive function to follow simple instructions and physically able to engage in sitting and standing exercises. (Chaovalit et al., 2021)

Exclusion Criteria:

* Joint contractures that interfere with bimanual tasks.
* History of upper limb orthopedic surgery
* Within the last half a year or botulinum toxin injections.
* Poor compliance with therapy.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Change in functional bimanual hand use as measured by the Able Hand Questionnaire (ABL) | Baseline and 8 weeks post-intervention
  The Able Hand Questionnaire (ABL) is a validated assessment tool used to evaluate functional use of both hands in daily activities for children with motor impairments. It consists of 21 items, each scored on a 3-point scale (easy, difficult, impossible), with higher scores indicating greater functional ability. The measure will be administered by a blinded assessor at baseline and after the 8-week intervention period to determine the change in bimanual performance between groups.

SECONDARY OUTCOMES:
Change in gross motor function classification (GMFCS level) | Baseline and 8 weeks post-intervention
  The Gross Motor Function Classification System (GMFCS) is a standardized tool for classifying motor function in children with cerebral palsy, ranging from Level I (least severe) to Level V (most severe). Classification will be performed at baseline and at the end of the 8-week intervention by a trained physiotherapist to monitor any changes in functional mobility classification. Although large changes in GMFCS level over short intervention periods are rare, the measure provides context for interpreting functional gains.
Caregiver-reported independence in daily activities | Baseline and 8 weeks post-intervention
  A structured caregiver questionnaire will be used to collect information on the child's ability to independently perform daily self-care tasks such as feeding, dressing, grooming, and play activities. The questionnaire will use a 3-point response scale (independent, requires assistance, dependent). This measure will be collected to assess perceived changes in independence associated with the intervention.
Adherence to home-based exercise program | Throughout the 8-week intervention period
  Adherence will be monitored through weekly caregiver logs documenting completion of assigned home-based activities. The number of completed sessions will be compared to the total prescribed sessions to calculate adherence percentage. This will help determine feasibility and engagement with the home component of the program.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No